CLINICAL TRIAL: NCT00686582
Title: An Open-Label Phase II Study to Evaluate Immunogenicity and Safety of a Single IMVAMUNE Booster Vaccination Two Years After the Last IMVAMUNE Vaccination in Former POX-MVA-005 Vaccinees
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: POX-MVA-023; EudraCT-No.2007-006297-28; DMID 08-0018
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-02

CONDITIONS: Smallpox
MeSH Terms: conditions — Smallpox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Initially Vaccinia Naive, 2 dose primed, 1 booster dose (Experimental): Group 1 Initially Vaccinia Naive Subjects 2 doses of MVA-BN in prior study (POX-MVA-005)
  1 booster dose of MVA-BN (POX-MVA-023) IMVAMUNE: 1x 10E8_TCID50
  Interventions: Biological: IMVAMUNE
- Initially Vaccinia Naive, 1 dose primed, 1 booster dose (Experimental): Group 2 Initially Vaccinia Naive Subjects 1 dose of MVA-BN and 1x Placebo in prior study (POX-MVA-005)
  1 booster dose of MVA-BN (POX-MVA-023) IMVAMUNE: 1x 10E8_TCID50
  Interventions: Biological: IMVAMUNE
- Vaccinia Experienced, boosted, blood draw only (Other): Group 4 Vaccinia Experienced
  1 booster dose of MVA-BN in prior study (POX-MVA-005) Blood draw, Screening Visit only (POX-MVA-023)
  Interventions: Procedure: Blood Draw Only

INTERVENTIONS:
Biological: IMVAMUNE — 1x 10E8_TCID50
  Arms: Initially Vaccinia Naive, 2 dose primed, 1 booster dose
Biological: IMVAMUNE — 1x 10E8_TCID50
  Arms: Initially Vaccinia Naive, 1 dose primed, 1 booster dose
Procedure: Blood Draw Only
  Arms: Vaccinia Experienced, boosted, blood draw only

SUMMARY:
The study was preformed to evaluate the persistence of antibodies following vaccination with MVA-BN and to assess the immunological memory response induced by a booster vaccination with MVA-BN in subjects two years after their participation in trial POX-MVA-005 (NCT00316524) in which they had received one or two doses of MVA-BN.

ELIGIBILITY:
Inclusion Criteria:

Groups 1 and 2 (first consenting 75 subjects in each group to be vaccinated)

* Male and female subjects having participated in Group 1 or 2 of the study POX-MVA-005 who completed the trial according to protocol.
* Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine or serum pregnancy test within 24 hours prior to vaccination.
* Women of childbearing potential must have used an acceptable method of contraception for 30 days prior to the vaccination, must agree to use an acceptable method of contraception during the study, and must not become pregnant for at least 28 days after the vaccination. A woman is considered of childbearing potential unless post-menopausal or surgically sterilized. (Acceptable contraception methods are restricted to abstinence, barrier contraceptives, intrauterine contraceptive devices or licensed hormonal products.)
* Read, signed and dated informed consent document after being advised of the risks and benefits of the study in a language understood by the subject signed, and prior to performance of any study specific procedure.
* Troponin I within normal institutional limits.
* White blood cells ≥ 2,500/mm3 and <= 11,000/mm3.
* Absolute neutrophil count within normal limits.
* Negative urine glucose by dipstick or urinalysis.
* Hemoglobin within the laboratory reference ranges (unless the investigator considers the deviation to be not clinically significant).
* Platelets 100 - 440/nL.
* Adequate renal function defined as:

  1. Serum creatinine without clinically significant findings.
  2. Urine protein <= 30 mg/dL or none or trace proteinuria (by urinalysis or dip stick).
* Adequate hepatic function defined as:

  1. Total bilirubin <= 1.5 x upper limit of normal (ULN) in the absence of other evidence of significant liver disease (healthy subjects without clinical disease; Morbus Meulengracht can be included).
  2. AST (SGOT), ALT (SGPT), alkaline phosphatase without clinically significant findings.
* Electrocardiogram (ECG) without clinically relevant abnormal findings (e.g. any kind of atrioventricular or intraventricular conditions or blocks such as complete left or right bundle branch block, AV node block, QTc or PR prolongation, premature atrial contractions or other atrial arrhythmia, sustained ventricular arrhythmia, two premature ventricular contractions (PVC) in a row, ST elevation consistent with ischemia).

Group 4 (all subjects) and Groups 1 and 2 (subjects N > 75): blood draw only

* Male and female subjects having participated in the study POX-MVA-005 who completed the trial according to protocol.
* Read, signed and dated informed consent document after being advised of the risks and benefits of the blood draw in a language understood by the subject signed, and prior to performance of the blood draw.

Exclusion Criteria:

Groups 1 and 2 (first consenting 75 subjects in each group to be vaccinated)

* Participation in another study with a smallpox vaccine after the POX-MVA-005 study.
* Pregnant or breast-feeding women.
* Uncontrolled serious infection i.e. not responding to antimicrobial therapy.
* History of any serious medical condition, which in the opinion of the investigator would compromise the safety of the subject.
* History of or active autoimmune disease. Persons with vitiligo or thyroid disease taking thyroid replacement are not excluded.
* Known or suspected impairment of immunologic function including, but not limited to, clinically significant liver disease; diabetes mellitus; moderate to severe kidney impairment.
* History of malignancy, other than squamous cell or basal cell skin cancer, unless there has been surgical excision that is considered to have achieved cure. Subjects with history of skin cancer must not be vaccinated at the previous site of cancer.
* History or clinical manifestation of clinically significant and severe hematological, renal, hepatic, pulmonary, central nervous, cardiovascular or gastrointestinal disorders.
* Clinically significant mental disorder not adequately controlled by medical treatment.
* Any condition which might interfere with study objectives or would limit the subject's ability to complete the study or to be compliant in the opinion of the investigator.
* History of coronary heart disease, myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, uncontrolled high blood pressure, or any other heart condition under the care of a doctor.
* History of an immediate family member (father, mother, brother, or sister) who died due to ischemic heart disease before age 50 years.
* Twenty percent or greater risk of developing a myocardial infarction or coronary death within the next 10 years using the National Cholesterol Education Program's risk assessment tool. (http://hin.nhlbi.nih.gov/atpiii/calculator.asp?usertype=prof).
* History of intravenous drug abuse.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. tris (hydroxymethyl)-amino methane, chicken embryo fibroblast proteins, aminoglycosides (gentamycin).
* History of any anaphylactic shock or severe allergic reaction requiring immediate treatment.
* Having received any vaccinations or planned vaccinations with a live vaccine within 30 days prior or after study vaccination.
* Having received any vaccinations or planned vaccinations with a killed vaccine within 14 days prior or after study vaccination.
* Chronic administration (defined as more than 14 days) of > 5 mg prednisone (or equivalent) per day or any other immune-modifying drugs during a period starting from three months prior to administration of the vaccine and ending at study conclusion (Visit 4).
* Post organ transplant subjects whether or not receiving chronic immunosuppressive therapy.
* Administration or planned administration of immunoglobulins and/or any blood products during a period starting from 3 months prior to administration of the vaccine and ending at study conclusion.
* Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceding administration of the study vaccine, or planned administration of such a drug during the study period.

Group 4 (all subjects) and Groups 1 and 2 (subjects N > 75): blood draw only

* Participation in another study with a smallpox vaccine after the POX-MVA-005 study.
* Any condition which might interfere with a blood draw.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 304 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Harrison Clinical Research Deutschland GmbH, München, Germany

REFERENCES:
- [Derived] Ilchmann H, Samy N, Reichhardt D, Schmidt D, Powell JD, Meyer TPH, Silbernagl G, Nichols R, Weidenthaler H, De Moerlooze L, Chen L, Chaplin P. One- and Two-Dose Vaccinations With Modified Vaccinia Ankara-Bavarian Nordic Induce Durable B-Cell Memory Responses Comparable to Replicating Smallpox Vaccines. J Infect Dis. 2023 May 12;227(10):1203-1213. doi: 10.1093/infdis/jiac455. PMID 36408618

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Initially Vaccinia Naive, 2 Dose Primed, 1 Booster Dose | Initially Vaccinia Naive, 1 Dose Primed, 1 Booster Dose | Vaccinia Experienced, Boosted, Blood Draw Only
Started (Blood Draw for Antibody Persistence 2 yrs after study POX-MVA-005) | 92 | 91 | 121
Booster Vaccination | 75 | 77 | 0
Completed (Active trial phase) | 74 | 77 | 121
Not Completed | 18 | 14 | 0

BASELINE CHARACTERISTICS:
Population: Persistence Set i.e. subjects previously vaccinated in study POX-MVA-005 with a blood draw at the screening visit of study POX-MVA-023
Groups:
- Total: Total of all reporting groups
Arm/Group | Initially Vaccinia Naive, 2 Dose Primed, 1 Booster Dose | Initially Vaccinia Naive, 1 Dose Primed, 1 Booster Dose | Vaccinia Experienced, Boosted, Blood Draw Only | Total
Number analyzed (Participants) | 92 | 91 | 121 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (5.8) | 27.7 (4.5) | 44.9 (6.6) | 34.6 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 55 | 67 | 172
  Male | 42 | 36 | 54 | 132
ELISA Long-Term Persistence [Geometric Mean (Full Range); unit: Titer] — Geometric Mean Titers (GMT) based on vaccinia-specific Enzyme-linked Immunosorbent Assay (ELISA) at the Screening Visit (2 years after one or two doses of MVA-BN in POX-MVA-005) are considered long-term immunogenicity outcomes from previous study. Titers below the detection limit are included with a value of '1'.
  Total Column: Pooled data is of limited relevance due to different precondition (naive vs experienced) / treatment (2 doses vs 1 dose of MVA-BN) in POX-MVA-005.
  Titer | 23.33 [1 to 1877] | 6.20 [1 to 262] | 134.65 [1 to 1103] | 31.52 [1 to 1877]
PRNT Long-Term Persistence [Geometric Mean (Full Range); unit: Titer] — Geometric Mean Titers (GMT) based on vaccinia-specific Plaque Reduction Neutralization Test (PRNT) at the Screening Visit (2 years after one or two doses of MVA-BN in POX-MVA-005) are considered long-term immunogenicity outcomes from previous study. Titers below the detection limit are included with a value of '1'.
  Total Column: Pooled data is of limited relevance due to different precondition (naive vs experienced) / treatment (2 doses vs 1 dose of MVA-BN) in POX-MVA-005.
  Titer | 1.26 [1 to 226] | 1.05 [1 to 67] | 10.28 [1 to 4382] | 2.75 [1 to 4382]

OUTCOME MEASURES:

1. Primary Outcome: Individual Peak Booster Rate by ELISA (Percentage of Participants)
Description: Booster rate based on vaccinia-specific Enzyme-linked Immunosorbent Assay (ELISA) is defined as the percentage of subjects with an appearance of antibody titers ≥ detection limit (50) for initially seronegative subjects, or an increase of the antibody titer compared to Baseline titer for initially seropositive subjects. Individual Peak booster rate is based on the maximum post-Baseline antibody titer within 4 weeks (measurements at Weeks 1, 2, and 4). Percentages based on number of subjects with data available.
Time Frame: within 4 weeks
Population: Full Analysis Set/ Booster Set i.e., all subjects having received a booster dose in POX-MVA-023. Thus, Group 4 is not included.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Initially Vaccinia Naive, 2 Dose Primed, 1 Booster Dose | Initially Vaccinia Naive, 1 Dose Primed, 1 Booster Dose
Number analyzed (Participants) | 75 | 77
percentage of subjects | 100.0 [95.2 to 100.0] | 100.0 [95.3 to 100.0]

2. Secondary Outcome: Booster Rate by ELISA (Percentage of Participants)
Description: Booster rate based on vaccinia-specific Enzyme-linked Immunosorbent Assay (ELISA) is defined as the percentage of subjects with an appearance of antibody titers ≥ detection limit (50) for initially seronegative subjects, or an increase of the antibody titer compared to Baseline titer for initially seropositive subjects. Percentages based on number of subjects with data available.
Time Frame: within 26 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Initially Vaccinia Naive, 2 Dose Primed, 1 Booster Dose | Initially Vaccinia Naive, 1 Dose Primed, 1 Booster Dose
Number analyzed (Participants) | 75 | 77
percentage of subjects
  Week 1 | 100.0 [95.2 to 100.0] | 98.7 [93.0 to 100.0]
  Week 2 | 100.0 [95.2 to 100.0] | 100.0 [95.3 to 100.0]
  Week 4: number analyzed (Participants) | 74 | 77
  Week 4 | 100.0 [95.1 to 100.0] | 100.0 [95.3 to 100.0]
  Week 26: number analyzed (Participants) | 71 | 77
  Week 26 | 98.6 [92.4 to 100.0] | 100.0 [95.3 to 100.0]

3. Secondary Outcome: ELISA GMT
Description: Geometric Mean Titers (GMT) based on vaccinia-specific Enzyme-linked Immunosorbent Assay (ELISA). Individual peak is defined as the maximum post-Baseline antibody titer within 4 weeks (measurements at Weeks 1, 2, and 4). Titers below the detection limit are included with a value of '1'.
Time Frame: within 26 weeks
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Initially Vaccinia Naive, 2 Dose Primed, 1 Booster Dose | Initially Vaccinia Naive, 1 Dose Primed, 1 Booster Dose
Number analyzed (Participants) | 75 | 77
Titer
  Screening | 24.23 [15.20 to 38.62] | 5.89 [3.63 to 9.57]
  Week 1 | 737.93 [597.37 to 911.58] | 490.33 [368.48 to 652.46]
  Week 2 | 1688.20 [1381.55 to 2062.91] | 1608.89 [1285.90 to 2013.00]
  Week 4 | 1255.21 [1029.02 to 1531.13] | 1210.59 [974.01 to 1504.62]
  Individual peak | 1821.57 [1496.13 to 2217.80] | 1723.74 [1376.87 to 2158.01]
  Week 26 | 461.78 [381.16 to 559.46] | 382.91 [301.66 to 486.03]

4. Secondary Outcome: Booster Rate by PRNT (Percentage of Participants)
Description: Booster rate based on vaccinia-specific Plaque Reduction Neutralization Test (PRNT) is defined as the percentage of subjects with an appearance of antibody titers ≥ detection limit (6) for initially seronegative subjects, or an increase of the antibody titer compared to Baseline titer for initially seropositive subjects.
  Individual Peak booster rate is based on the maximum post-Baseline antibody titer within 4 weeks (measurements at Weeks 1, 2, and 4).
  Percentages based on number of subjects with data available.
Time Frame: within 26 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Initially Vaccinia Naive, 2 Dose Primed, 1 Booster Dose | Initially Vaccinia Naive, 1 Dose Primed, 1 Booster Dose
Number analyzed (Participants) | 75 | 77
percentage of subjects
  Week 1 | 92.0 [83.4 to 97.0] | 85.7 [75.9 to 92.6]
  Week 2 | 98.7 [92.8 to 100.0] | 96.1 [89.0 to 99.2]
  Week 4: number analyzed (Participants) | 74 | 77
  Week 4 | 94.6 [86.7 to 98.5] | 90.9 [82.2 to 96.3]
  Individual peak | 98.7 [92.8 to 100.0] | 98.7 [93.0 to 100.0]
  Week 26: number analyzed (Participants) | 71 | 77
  Week 26 | 88.7 [79.0 to 95.0] | 76.6 [65.6 to 85.5]

5. Secondary Outcome: PRNT GMT
Description: Geometric Mean Titers (GMT) based on vaccinia-specific Plaque Reduction Neutralization Test (PRNT). Individual peak is defined as the maximum post-Baseline antibody titer within 4 weeks (measurements at Weeks 1, 2, and 4). Titers below the detection limit are included with a value of '1'.
Time Frame: within 26 weeks
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Initially Vaccinia Naive, 2 Dose Primed, 1 Booster Dose | Initially Vaccinia Naive, 1 Dose Primed, 1 Booster Dose
Number analyzed (Participants) | 75 | 77
Titer
  Screening | 1.23 [0.99 to 1.52] | 1.06 [0.95 to 1.18]
  Week 1 | 53.61 [37.05 to 77.59] | 28.58 [18.56 to 43.99]
  Week 2 | 125.26 [89.51 to 175.27] | 80.69 [54.37 to 119.75]
  Week 4 | 64.26 [43.19 to 95.61] | 48.96 [31.72 to 75.57]
  Individual Peak | 165.97 [124.21 to 221.77] | 116.79 [82.42 to 165.49]
  Week 26 | 49.29 [32.40 to 74.98] | 25.62 [15.84 to 41.44]

6. Secondary Outcome: Correlation PRNT vs ELISA Titers
Description: Pearson Correlation Coefficient between the log10 transformed PRNT titers and the log10 transformed ELISA titers
Time Frame: within 26 weeks
Population: as for outcome 1
Measure: Number; unit: Pearson correlation coefficient
Arm/Group | Initially Vaccinia Naive, 2 Dose Primed, 1 Booster Dose | Initially Vaccinia Naive, 1 Dose Primed, 1 Booster Dose
Number analyzed (Participants) | 75 | 77
Pearson correlation coefficient
  Week 1 | 0.591 | 0.690
  Week 2 | 0.491 | 0.655
  Week 4 | 0.476 | 0.592
  Week 26 | 0.568 | 0.550

7. Secondary Outcome: Number of Participants With Related Serious Adverse Events
Description: Number of participants with Serious Adverse Events (SAEs) probably, possibly or definitely related to the trial vaccine
Time Frame: within 26 weeks
Population: Full Analysis Set/ Booster Set i.e., all subjects having received a booster dose in POX-MVA-023. Subjects from Group 4 had a blood draw at Screening only, did not receive a booster dose and adverse events were not monitored/assessed for this group.
Measure: Count of Participants; unit: Participants
Arm/Group | Initially Vaccinia Naive, 2 Dose Primed, 1 Booster Dose | Initially Vaccinia Naive, 1 Dose Primed, 1 Booster Dose
Number analyzed (Participants) | 75 | 77
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With Unsolicited Non-serious Adverse Events
Description: Number of participants with any, grade >=3, and related non-serious unsolicited adverse events
Time Frame: within 29 days after any vaccination
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Initially Vaccinia Naive, 2 Dose Primed, 1 Booster Dose | Initially Vaccinia Naive, 1 Dose Primed, 1 Booster Dose
Number analyzed (Participants) | 75 | 77
Participants
  Any event | 40 | 38
  Any event with intensity >= Grade 3 | 4 | 5
  Any event assessed as related to vaccine | 11 | 9

9. Secondary Outcome: Number of Participants With Related Grade >= 3 Unsolicited Adverse Events
Description: Number of participants with Grade >=3 Unsolicited Adverse Event probably, possibly, or definitely related to the study vaccine
Time Frame: within 29 days after vaccination
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Initially Vaccinia Naive, 2 Dose Primed, 1 Booster Dose | Initially Vaccinia Naive, 1 Dose Primed, 1 Booster Dose
Number analyzed (Participants) | 75 | 77
Participants | 1 | 0

10. Secondary Outcome: Number of Participants With Solicited Local Adverse Events
Description: Number of participants with and intensity of solicited local AEs (pain, erythema, swelling, induration, and pruritis). Percentages based on subjects with a completed diary card.
Time Frame: within 8 days after vaccination
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Initially Vaccinia Naive, 2 Dose Primed, 1 Booster Dose | Initially Vaccinia Naive, 1 Dose Primed, 1 Booster Dose
Number analyzed (Participants) | 75 | 77
Participants
  Pain: Any | 58 | 64
  Pain: Grade >=3 | 1 | 3
  Erythema: Any | 60 | 65
  Erythema: Grade >=3 | 0 | 2
  Swelling: Any | 51 | 48
  Swelling: Grade >=3 | 0 | 2
  Induration: Any | 58 | 58
  Induration: Grade >=3 | 0 | 1
  Pruritis: Any | 30 | 36
  Pruritis: Grade >=3 | 1 | 0

11. Secondary Outcome: Number of Participants With Solicited General Adverse Events
Description: Number of participants with solicited general AEs (body temperature increased, headache, myalgia, nausea, and fatigue): Intensity and relationship to vaccination. Percentages based on subjects with a completed diary card.
Time Frame: within 8 days after vaccination
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Initially Vaccinia Naive, 2 Dose Primed, 1 Booster Dose | Initially Vaccinia Naive, 1 Dose Primed, 1 Booster Dose
Number analyzed (Participants) | 75 | 77
Participants
  Body temperature increased: Any | 3 | 4
  Body temperature increased: Grade >=3 | 0 | 0
  Body temperature increased: Related Grade >=3 | 0 | 0
  Headache: Any | 19 | 25
  Headache: Grade >=3 | 2 | 1
  Headache: Related Grade >=3 | 1 | 1
  Myalgia: Any | 17 | 19
  Myalgia: Grade >=3 | 1 | 1
  Myalgia: Related Grade >=3 | 1 | 0
  Nausea: Any | 6 | 12
  Nausea: Grade >=3 | 0 | 0
  Nausea: Related Grade >=3 | 0 | 0
  Fatigue: Any | 22 | 27
  Fatigue: Grade >=3 | 2 | 0
  Fatigue: Related Grade >=3 | 2 | 0

ADVERSE EVENTS:
Time Frame: 7 months
Description: AEs only collected for subjects that received a booster dose in POX-MVA-023. Subjects from Group 4 had a blood draw at Screening only, did not receive a booster dose and adverse events were not monitored/assessed for this group.
Arm/Group | Initially Vaccinia Naive, 2 Dose Primed, 1 Booster Dose | Initially Vaccinia Naive, 1 Dose Primed, 1 Booster Dose
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/77
Serious Adverse Events (participants affected / at risk) | 2/75 | 0/77
Other Adverse Events (participants affected / at risk) | 35/75 | 25/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initially Vaccinia Naive, 2 Dose Primed, 1 Booster Dose (N=75) | Initially Vaccinia Naive, 1 Dose Primed, 1 Booster Dose (N=77)
Gastroenteritis (Infections and infestations) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Initially Vaccinia Naive, 2 Dose Primed, 1 Booster Dose (N=75) | Initially Vaccinia Naive, 1 Dose Primed, 1 Booster Dose (N=77)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 3
Palpitations (Cardiac disorders) | 2 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 2
Toothache (Gastrointestinal disorders) | 2 | 0
Chills (General disorders) | 0 | 2
Injection site irritation (General disorders) | 2 | 0
Injection site warmth (General disorders) | 3 | 3
Nasopharyngitis (Infections and infestations) | 20 | 9
Limb injury (Injury, poisoning and procedural complications) | 0 | 2
Headache (Nervous system disorders) | 5 | 7
Migraine (Nervous system disorders) | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes